CLINICAL TRIAL: NCT05341492
Title: A Single-arm, Open, Exploratory Clinical Study Evaluating the Safety and Efficacy of EGFR/B7H3 CAR-T in Patients With EGFR/ B7H3-positive Advanced Solid Tumors (Lung and Triple-negative Breast Cancer)
Brief Title: EGFR/B7H3 CAR-T on Lung Cancer and Triple Negative Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZBGCART-016
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: EGFR/ B7H3-positive Advanced Lung Cancer; EGFR/ B7H3-positive Advanced Triple-negative Breast Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Patients will receive 2*10e6/kgCAR-T cells.
  Interventions: Biological: EGFR/B7H3 CAR-T

INTERVENTIONS:
Biological: EGFR/B7H3 CAR-T — 2 × 10^6/kg CAR-T cells,For subjects with body weight greater than 60 kg, the number of cells can only be calculated according to 60 kg of body weight.

SUMMARY:
This study is a single-arm, open, exploratory clinical study to evaluate the safety and efficacy of EGFR/B7H3 CAR-T in patients with EGFR/ B7H3-positive advanced solid tumors (lung cancer and triple-negative breast cancer)

ELIGIBILITY:
Inclusion Criteria:

* 1.All subjects or legal guardians must sign the informed consent form approved by the ethics committee in writing before starting any screening procedure;
* 2.18 Years to 75 Years, Histologically or cytologically confirmed Routine treatment of patients with advanced lung cancer and triple-negative breast cancer(Including TKI treatment failure patients);
* 3.EGFR/B7H3 expression was confirmed positive in tumor site by immunohistochemical test within 3 months before signing the informed consent form;
* 4.According to RECIST version 1.1 of solid tumor efficacy evaluation criteria, there should be at least one measurable lesion during screening period (results are available within one month prior to screening period) ;
* 5.Expected survival time ≥ 12 weeks;
* 6.The Eastern oncology group strength status score (ECOG) was 0-1;
* 7.Adequate organ function: alanine aminotransferase, aspartate aminotransferase (ALT, AST) < 3 times of normal value, total bilirubin (TBiL) < 1.5 times of normal value, serum creatinine (SCr) < 1.5 times of normal value;
* 8.The hemodynamics determined by echocardiography or multichannel radionuclide angiography(MUGA) are stable and the left ventricular ejection fraction (LVEF)≥50%;
* 9.Have sufficient bone marrow reserves (subjects can meet this requirement through blood transfusion), defined as: The number of white blood cells should not be less than 1 × 10^9/L;Platelet≥100 x 10^9/L; Hemoglobin ≥100 g/L;
* 10.Women of childbearing age and all male subjects must agree to use effective contraceptive methods for at least 52 weeks after EGFR CAR-T infusion, and until two consecutive PCR tests show that CAR-T cells are no longer present in the body.

Exclusion Criteria:

* 1.Uncontrolled hypertension (> 160/95), unstable coronary artery disease confirmed by uncontrolled arrhythmia, unstable angina pectoris, decompensated congestive heart failure (> New York Heart Association Class II), or myocardial infarction within 6 months prior to cell infusion;
* 2.Patients with severe liver and kidney dysfunction or consciousness disorder;
* 3.Patients who received antitumor chemotherapy other than lymphocyte clearance chemotherapy within 14 days prior to CAR T infusion;
* 4.Patients who received other study drugs within 14 days prior to infusion;
* 5. Patients treated with radiotherapy or TKI within 2 weeks prior to infusion;
* 6. Patients with active hepatitis B: HBV DNA>1000IU/mL;
* 7. HIV antibody, hepatitis C antibody, treponema pallidum antibody positive patients;
* 8. Sputum smears and patients who test positive for T cells of tuberculosis infection
* 9.Patients with interstitial lung disease or pneumonia;
* 10.patients with uncontrolled acute life-threatening bacterial, viral or fungal infection (e.g. positive blood culture ≤72 hours prior to infusion);
* 11.Patients with central nervous primary tumor or central metastasis solid tumor (patients with stable treatment for more than 4 weeks after brain metastasis or patients with asymptomatic brain metastasis without treatment are excluded from this range), and patients with pericardial metastasis accompanied by large pericardial effusion.
* 12.Patients with a prior or concurrent second tumor, except in the following cases:

  * Adequately treated basal cell or squamous cell carcinoma (adequate wound healing required prior to enrollment);
  * Carcinoma in situ of cervical or breast cancer with no signs of recurrence for at least 3 years prior to study after curative treatment;
  * The primary malignancy has been completely resected and in complete remission for ≥5 years.
* 13.Pregnant or lactating women;
* 14.Patients who have a history of or currently have T-cell tumors;
* 15. have active neuroautoimmune or inflammatory disorders (e.g. Guillian-Barre syndrome, AMyotrophic lateral sclerosis);
* 16.Other conditions, such as compliance, that the investigator considers should not be included in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
Safety by Common Terminology Criteria for Adverse Events (CTCAE) V5.0 | In CAR-T cells infusion, up to 52 weeks.
  The type, frequency, severity, and duration of adverse events as a result of EGFR/B7H3 CAR-T cells infusion will be summarized

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | In CAR-T cells infusion, up to 52 weeks.
  Per Response Evaluation Criteria in Solid Tumours (RECIST 1.1) assessed by MRI or CT. ORR is the percentage of patients at Complete Response (CR) or Partial Response (PR) (according to independent review), prior to progression or further anti-cancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Luo min, PhD, Study Chair — Guangzhou Bio-gene Technology Co., Ltd
Locations (1):
- Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No